CLINICAL TRIAL: NCT02968628
Title: Effect of Maternal Diabetes on Brain Development, as Measured by Neonatal Electroencephalogram (EEG)
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: RSRB00061973
Record Dates: First submitted 2016-08-26; First posted 2016-11-18 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes in Pregnancy; Diabetes, Gestational; Infant, Newborn, Diseases; Perinatal Disorders of Growth and Development
MeSH Terms: conditions — Diabetes, Gestational; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Infants of Diabetic Mothers: Cases: Neonates born at or over 35 weeks gestation whose mother's were recommended to receive medication for diabetes during pregnancy. This includes pre-gestational and gestational diabetics.
  Interventions:
  1. Video Electroencephalogram (EEG)
  2. Point-of Care Blood Sugar Testing
  3. Medical Record Data Extraction
  4. Maternal Questionnaire
  Interventions: Other: Video Electroencephalogram (EEG); Other: Point-of Care Blood Sugar Testing; Other: Medical Record Data Extraction; Other: Maternal Questionnaire
- Controls: Controls: Neonates born at or over 35 weeks gestation whose mother's had normal glycemic control testing during pregnancy.
  Interventions:
  1. Video Electroencephalogram (EEG)
  2. Point-of Care Blood Sugar Testing
  3. Medical Record Data Extraction
  4. Maternal Questionnaire
  Interventions: Other: Video Electroencephalogram (EEG); Other: Point-of Care Blood Sugar Testing; Other: Medical Record Data Extraction; Other: Maternal Questionnaire

INTERVENTIONS:
Other: Video Electroencephalogram (EEG) — Single neonatal video EEG at 24 hrs to 5 days of life during birth hospitalization. Neonatal scalp leads, respiratory and nasal leads. Approximately 60 minute recording.
Other: Point-of Care Blood Sugar Testing — One-time heel-stick point-of-care blood sugar testing at time of EEG.
Other: Medical Record Data Extraction — Medical record data extraction from both maternal obstetric and neonatal medical record for variables known to impact EEG and neurodevelopmental outcomes.
Other: Maternal Questionnaire — One-time maternal questionnaire related to smoking practices, ETOH consumption, level of education, and body mass index.

SUMMARY:
Alterations in the intrauterine environment can have profound effects on fetal development. Diabetes during gestation results in multiple deleterious short-term outcome differences, and is correlated with long-term developmental deficits. Multiple studies, in neonates through school-aged children, have demonstrated differences in language, attention and psychomotor development in offspring of diabetic pregnancies. Neonatal EEG is a promising and non-invasive tool for assessment of abnormal brain development or "dysmaturity" in this population. Multiple conventional EEG (cEEG) and amplitude-integrated EEG (aEEG) parameters change predictably with advancing gestational development and have been used to differentiate between at risk groups in neonatal studies.

The investigators hypothesize that neonatal EEG can identify brain dysmaturity in infants of diabetic mothers (IDMs) compared to gestational-age matched controls. The primary aim is documentation of brain dysmaturity in IDMs using cEEG. The secondary aim is establishment of aEEG as a more accessible tool to quantify the effects of maternal diabetes on neonatal brain development.

The investigators will conduct a pilot study comparing cEEG and aEEG parameters of cases to gestational-age matched controls. Cases will be IDM neonates of at least 35 weeks' gestation whose mothers were recommended treatment with either insulin or an oral glycemic agent. Video EEG recording will be planned for approximately 60 minutes and obtained between 24 hours and 5 days of life during birth hospitalization. Additional data will be extracted from maternal and neonatal medical records and a maternal questionnaire.

In addition to evaluating the measures of cEEG and aEEG, this project will establish a research cohort. A subsequent study involving developmental evaluations will allow for correlation of EEG results with long-term outcomes. The ability to identify those at risk at birth would provide the opportunity to intervene in order to mitigate outcome differences, particularly in language development. More significantly, we hope to establish neonatal CNS outcome measures for future diabetic pregnancy intervention studies. .

ELIGIBILITY:
Inclusion Criteria:

* >/= 35 weeks post-menstrual age at delivery
* Dating by, or consistent with, 1st trimester ultrasound
* Mother able to communicate in oral and written English
* Available maternal obstetric record and medication history
* Singleton gestation
* Delivery at URMC attended by obstetric staff

Exclusion Criteria:

Maternal Exclusion Criteria:

* Diagnosis by obstetrician of intrauterine growth restriction (IUGR)
* Documentation in medical record of daily maternal cigarette smoking during 2nd or 3rd trimester
* Chronic maternal sedative or opiate use (>weekly use)
* Recreational opiate use or addiction
* Cocaine or amphetamine use during pregnancy
* ETOH abuse or concern for abuse during pregnancy (>weekly use)
* Other maternal conditions that may compromise fetus
* Psychiatric medications beyond isolated SSRI use
* Anti-epileptic drugs (AEDs) during gestation
* Magnesium exposure within 3 days of delivery

Neonatal Exclusion Criteria:

* Blood gas pH of less than 7.1, if obtained (cord or any prior to EEG)
* Apgar less than 8 at 5 min
* CNS malformations, seizures, subgaleal or intracranial bleeds
* Cardiac anomalies except asymptomatic small-moderate VSD, ASD, or PDA
* Clinically significant malformations or chromosomal anomalies
* Small-for-gestational age (<10th % on Fenton growth curve)
* Respiratory distress ever requiring intubation or requiring CPAP support > 48 hours
* Hemodynamic instability requiring use of pressors or >2 bolus
* Culture positive sepsis
* Clinical concern for meningitis or encephalopathy
* Sedation medication or other conditions/medications affecting CNS function
* Clinically obtained total bilirubin more than 15 on day of EEG
* Scalp injury preventing placement of EEG leads
* Point-of-care testing (POCT) glucose <45 at time of EEG

Ages: 24 Hours to 120 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be a convenience sample, comprised of singleton neonates born at or after 35 weeks post-menstrual age at the University of Rochester Medical Center (URMC). Cases will be infants of mothers with either a diagnoses of pre-gestational diabetes or gestational diabetes whose provider recommends treatment with insulin or oral glycemic agents. Controls will be neonates whose mothers had normal glucose testing during gestation and pre-pregnancy BMI of <30. All subjects will be otherwise healthy, as defined by the exclusion criteria. There is no intended racial, ethnic or gender distribution of these neonates.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum Interburst Interval on cEEG | Single EEG between 24 hours of life and 5 days of life
Lower Margin Amplitude on aEEG | Single EEG between 24 hours of life and 5 days of life

SECONDARY OUTCOMES:
Number of Delta Brushes on cEEG | Single EEG between 24 hours of life and 5 days of life
Bandwidth on aEEG | Single EEG between 24 hours of life and 5 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Price, MD, Principal Investigator — University of Rochester; Ronnie Guillet, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No